CLINICAL TRIAL: NCT05654935
Title: Telerobotic Ultrasound for Carotid Imaging - Feasibility Study
Status: Withdrawn | Type: Observational
Why Stopped: Failure to procure funding and technical logistics
Sponsor: Rush University Medical Center (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Rami Doukky, Professor of Medicine, Preventive Medicine, and Radiology, Rush University Medical Center; Interim Chief Division of Cardiology, John H. Stroger, Jr. Hospital of Cook County, Rush University Medical Center
Other Study IDs: 13090301-IRB01
Record Dates: First submitted 2022-12-08; First posted 2022-12-16 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Carotid Artery Disease; Atherosclerosis; Atheromatous Plaques; Arteriosclerosis; Vascular Disease; Arterial Occlusive Diseases; Stroke; Cardiac Death; Myocardial Infarction; Coronary Artery Disease; Cardiovascular Disease; Coronary Disease; Coronary Arteriosclerosis; Carotid Arteriosclerosis; Myocardial Ischemia; Heart Diseases; Cerebrovascular Disorders; Peripheral Vascular Disease; Cerebrovascular Accident; Cerebral Infarction
MeSH Terms: conditions — Carotid Artery Diseases; Atherosclerosis; Plaque, Atherosclerotic; Arteriosclerosis; Vascular Diseases; Arterial Occlusive Diseases; Stroke; Death; Myocardial Infarction; Coronary Artery Disease; Cardiovascular Diseases; Coronary Disease; Myocardial Ischemia; Heart Diseases; Cerebrovascular Disorders; Peripheral Vascular Diseases; Cerebral Infarction | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cohort A: Includes 26 healthy volunteers >18 years of age without history of stroke or transient ischemic attack, coronary artery disease (prior myocardial infarction, typical angina, prior percutaneous coronary revascularization, and prior coronary bypass graft surgery), and peripheral arterial disease (claudication, peripheral arterial revascularization stenting of bypass surgery). Subjects will be recruited using advertisement flyers and emails.
  Interventions: Radiation: Ultrasound for Carotid Arteries; Radiation: Telerobotic Ultrasound for Carotid Arteries
- Cohort B: Includes 100 subjects ≥ 60 years of age without known carotid artery disease. These subjects will be recruited from patients scheduled to receive a clinically indicated cardiac stress test or echocardiogram in the noninvasive cardiac testing area at Rush University Medical Center (Chicago, IL).
  Interventions: Radiation: Ultrasound for Carotid Arteries; Radiation: Telerobotic Ultrasound for Carotid Arteries

INTERVENTIONS:
Radiation: Ultrasound for Carotid Arteries — Cohort A: each subject will undergo two manual ultrasound image acquisitions by two different registered vascular sonographers who will be blinded to one another's images and findings.
  Cohort B: each subject in Cohort B will undergo one manual ultrasound acquisition conducted at Rush University Medical Center.
  Other Names: Carotid Ultrasound; Ultrasonography
Radiation: Telerobotic Ultrasound for Carotid Arteries — Cohort A: each subject will undergo two separate telerobotic acquisitions, in which the robotic arm will be controlled by two separate sonographers from Mount Sinai Medical Center (New York, NY). The sonographers controlling the robotic arm will be blinded to one another's images and to the images from the manual acquisition.
  Cohort B: each subject will undergo one telerobotic ultrasound (in random sequence with the manual acquisition also performed for this cohort) acquired by a separate technologist than the technologist that acquired the subject's manual ultrasound. This acquisition will be conducted at Rush University Medical Center by a technologist blinded to the images of the manual acquisition technologist. Robotic acquisition will be manipulated from a different building at Rush University Medical Center using a broadband cellular internet signal (rather than the institutional intranet).
  Other Names: Carotid Ultrasound; Telerobotic Ultrasonography

SUMMARY:
In this proposal, the investigators will demonstrate the feasibility and noninferiority of telerobotic ultrasonography as compared to traditional manual acquisition in performing a limited carotid Duplex examination and in carotid plaque detection.

DETAILED DESCRIPTION:
BACKGROUND

Ultrasonography is an inexpensive, noninvasive, radiation-free diagnostic tool that is indispensable in modern medicine. Carotid intima-media thickness (IMT) and carotid atherosclerotic plaque detection have been powerful screening tools for identifying patients at risk for cardiovascular events; including myocardial infarction, cardiac death, and stroke. The need for trained sonographers by the patient side to perform quality ultrasound studies has limited the accessibility to this imaging tool, both in terms of location and time of day. Robotic arms controlled remotely over the internet, by trained sonographers, can potentially provide easier and more ubiquitous access to ultrasonography in and outside traditional medical facilities, including remote villages in underdeveloped countries, disaster areas, battle zones, etc. In this proposal, the investigators will demonstrate the feasibility and noninferiority of telerobotic ultrasonography as compared to traditional manual acquisition in performing a limited carotid Duplex examination and in carotid plaque detection.

HYPOTHESIS:

Telerobotic ultrasound performed by an experienced sonographer over the Internet produces diagnostic images with quality similar to manual conventional imaging.

AIMS:

1. Telerobotic ultrasonography produces diagnostic images of the carotid arteries at a rate that is non-inferior to those obtained using standard manual acquisition.
2. Telerobotic ultrasonography can detect carotid atherosclerotic plaques at a rate that is non-inferior to the gold standard of manual acquisition.

IMPLICATIONS:

Realizing our study aims could mark a new era in ultrasonography. There are wide applications for telerobotic carotid ultrasonography in atherosclerosis screening. Furthermore, establishing the noninferiority of telerobotic carotid ultrasonography acquisition will provide a rationale for further studies in telerobotic ultrasonography, including echocardiography. This in turn has even wider clinical applications such as emergency studies in hospitals during weekends and after-hours. In addition, this could pave the way for use in disaster areas and battle zones where expert sonographers may not be available on-site.

ELIGIBILITY:
Inclusion Criteria for Cohort A

* Healthy volunteer
* >18 years of age
* Signed informed consent

Exclusion criteria for Cohort A include:

* Prior stroke or transient ischemic attack
* Prior heart attack.
* Prior angioplasty/stent of the heart artries
* Prior bypass surgery of the heart
* Known history of peripheral arterial disease claudication Peripheral arterial revascularization
* known history of carotid artery stenosis

Exclusion criteria for Cohort B include:

* known history of carotid artery stenosis
* known history carotid artery dissection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study aims will be realized in two separate populations:
  1. Cohort A: Includes 26 healthy volunteers >18 years of age.
  2. Cohort B: Includes 100 patients ≥ 60 years of age without known carotid artery disease. These patients will be recruited from patients scheduled to receive a clinically indicated cardiac stress test or echocardiogram in the noninvasive cardiac testing area at Rush University Medical Center (Chicago, IL). Patients will be approached regarding their interest in participating in the proposed investigation while waiting for their
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-03-26 (Actual); Primary Completion 2015-03-25 (Actual); Study Completion 2016-03-25 (Actual)

PRIMARY OUTCOMES:
Diagnostic Quality of Telerobotic Ultrasound. | 3 months
  Gray scale examination of the right and left carotid arteries in 3 views: short axis view of the common carotid artery, long axis view of carotid bifurcation, and short axis view post bifurcation. Images will be analyzed for:
  1. Diagnostic image quality (diagnostic vs. non-diagnostic quality) by 2 reviewers blinded to image acquisition modality (manual vs. telerobotic).
  2. Image quality graded on a scale from 1 to 4 by the same two reviewers as 1) poor/non-diagnostic; 2) fair; 3) acceptable; 4) good/excellent.
  Evaluation for diagnostic quality will be performed by two independent observers who will be blinded to the modality of image acquisition. Disagreement between observers will be resolved by a third blinded observer.

SECONDARY OUTCOMES:
Carotid Intima-Media Thickness (CIMT) Measurement | 3 months
  The subjects will be evaluated for the presence or absence of carotid artery atherosclerotic plaques. Each carotid artery (left and right) will be treated as an independent subject. Agreement analysis in the diagnosis of carotid artery plaques, between manual and telerobotic acquisition, will be performed. Identification of carotid artery plaques will be performed by two independent observers. Disagreements will be resolved by a third blinded observer.
Subject Experience with Manual vs. Telerobotic Ultrasound | 3 months
  Subject experience with each imaging technique (manual vs. telerobotic) will be determined by a simple questionnaire, as follows:
  1. How did the subject feel during the examination? Comfortable; fairly comfortable; somewhat uncomfortable; very uncomfortable.
  2. Would the subject have this test again in the future? Definitely, probably; probably not, definitely not.